CLINICAL TRIAL: NCT02589665
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Parallel, Placebo-Controlled Study of LY3074828 in Subjects With Moderate to Severe Ulcerative Colitis
Brief Title: A Study of Mirikizumab (LY3074828) in Participants With Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15829; I6T-MC-AMAC (Other: Eli Lilly and Company); 2015-003123-57 (EudraCT Number)
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Results first posted 2020-05-29 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Ulcerative Colitis
Keywords: IL-23 antibody
MeSH Terms: conditions — Colitis, Ulcerative | interventions — mirikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- 50 mg Mirikizumab IV Q4W (Induction) (Experimental): 50 mg mirikizumab administered every 4 weeks (Q4W) intravenously (IV) during the induction period. Participants who do not have a clinical response may choose to participate in the unblinded study extension period.
  Interventions: Drug: Mirikizumab
- 200 mg Mirikizumab IV Q4W (induction) (Experimental): 200 mg mirikizumab administered every 4 weeks (Q4W) intravenously (IV) during the induction period.
  Participants who do not have a clinical response may choose to participate in the unblinded study extension period.
  Interventions: Drug: Mirikizumab
- 600 mg Mirikizumab IV Q4W (Induction) (Experimental): 600 mg mirikizumab administered every 4 weeks (Q4W) intravenously (IV) during the induction period.
  Participants who do not have a clinical response may choose to participate in the unblinded study extension period.
  Interventions: Drug: Mirikizumab
- Placebo IV Q4W (Induction) (Placebo Comparator): Placebo administered every 4 weeks (Q4W) intravenously (IV) during the induction period.
  Interventions: Drug: Placebo
- 200 mg Mirikizumab SC Q4W (Maintenance) (Experimental): Induction mirikizumab responders were re-randomized: 200 mg mirikizumab administered subcutaneously (SC) Q4W during the maintenance period.
  Interventions: Drug: Mirikizumab
- 200 mg Mirikizumab SC Q12W (Maintenance) (Experimental): Induction mirikizumab responders were re-randomized: 200 mg mirikizumab administered subcutaneously (SC) once every 12 weeks (Q12W) during the maintenance period.
  Interventions: Drug: Mirikizumab
- Placebo SC Q4W (Maintenance) (Placebo Comparator): Induction placebo responders: Placebo administered subcutaneously (SC) Q4W during the maintenance period.
  Interventions: Drug: Placebo
- 600mg Mirikizumab IV Q4W Extension Open-Label (Experimental): Induction non-responders: 600 mg mirikizumab administered intravenously (IV) once every 4 weeks (Q4W) during the Extension Open-Label.
  Interventions: Drug: Mirikizumab
- 1000mg Mirikizumab IV Q4W Extension Open-Label (Experimental): Induction non-responders: 1000 mg mirikizumab administered intravenously (IV) once every 4 weeks (Q4W) during the Extension Open-Label.
  Interventions: Drug: Mirikizumab
- 200mg Mirikizumab SC Q4W Extension Open-Label (Experimental): Extension Induction responders: 200 mg mirikizumab administered subcutaneously (SC) once every 4 weeks (Q4W) during the Extension Open-Label
  Interventions: Drug: Mirikizumab

INTERVENTIONS:
Drug: Mirikizumab
  Other Names: LY3074828
  Arms: 1000mg Mirikizumab IV Q4W Extension Open-Label; 200 mg Mirikizumab IV Q4W (induction); 200 mg Mirikizumab SC Q12W (Maintenance); 200 mg Mirikizumab SC Q4W (Maintenance); 200mg Mirikizumab SC Q4W Extension Open-Label; 50 mg Mirikizumab IV Q4W (Induction); 600 mg Mirikizumab IV Q4W (Induction); 600mg Mirikizumab IV Q4W Extension Open-Label
Drug: Placebo
  Arms: Placebo IV Q4W (Induction); Placebo SC Q4W (Maintenance)

SUMMARY:
The main purpose of this study is to test the hypothesis that treatment with mirikizumab is superior to placebo in providing clinical benefit to participants with moderate to severe ulcerative colitis (UC). This study will also investigate how the body processes the drug.

ELIGIBILITY:
Inclusion Criteria:

* Have moderate to severe active UC as defined by a Mayo score of 6 to 12 with an endoscopic subscore ≥2 within 14 days before the first dose of study treatment (note: a partial Mayo score of at least 4 and other eligibility criteria must have been met before endoscopy is performed as a study procedure)
* Have evidence of UC extending proximal to the rectum (≥15 centimeters [cm] of involved colon)
* Up-to-date colorectal cancer surveillance (performed according to local standard), for subjects with family history of colorectal cancer, personal history of increased colorectal cancer risk, age >50 years, or other known risk factor
* Participants must either: be naive to biologic therapy (eg, tumor necrosis factor [TNF] antagonists or vedolizumab) and have at least 1 of the following: inadequate response or failure to tolerate current treatment with oral or intravenous corticosteroids or immunomodulators (6-mercaptopurine or azathioprine) or history of corticosteroid dependence (an inability to successfully taper corticosteroids without return of UC) OR have received treatment with 1 or more biologic agents (eg, TNF antagonists or vedolizumab) at doses approved for the treatment of UC with documented history of failure to respond to or tolerate such treatment

Exclusion Criteria:

* Have been diagnosed with indeterminate colitis, proctitis (distal disease involving the rectum only; less than 15 cm from the anal verge) or Crohn's Disease
* Have had surgery for treatment of UC or are likely to require surgery for UC during the study
* Have received any of the following for treatment of UC: cyclosporine or thalidomide within 30 days of screening, corticosteroid enemas, corticosteroid suppositories, or topical treatment with 5-aminosalicyclic acid within 30 days of screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2019-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (71):
- United States (11):
  - Precision Research Institute, LLC, Chula Vista, California
  - University of California - San Diego, La Jolla, California
  - Inland Empire Liver Foundation, Rialto, California
  - Borland Groover Clinic, Jacksonville, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Delta Research Partners LLC, Monroe, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Minnesota Gastroenterology, P.A., Plymouth, Minnesota
  - Columbia University Medical Center, New York, New York
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Care Access Research - Salt Lake City, Salt Lake City, Utah
- Australia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Concord
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fitzroy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Brisbane
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woolloongabba
- Belgium (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ghent
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leuven
- Canada (4):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Calgary
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Montreal
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal
- Czechia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hradec Králové
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Prague
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Praha 4 Kralove
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Svendborg, Denmark
- France (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clichy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint-Priest-en-Jarez
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vandœuvre-lès-Nancy
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tbilisi, Georgia
- Hungary (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Békéscsaba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szeged
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szekszárd
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vác
- Japan (18):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bunkyō City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Chūōku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagoshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kamakura-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Kasugai-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kawasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Mitaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Nishinomiya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Sakura
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shinjuku-ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Takasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Toyama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toyota-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Tsu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Yokohama
- Lithuania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaunas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vilnius
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chisinau, Moldova
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam, Netherlands
- Poland (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydgoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Elblag
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Katowice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rzeszów
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sopot
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest, Romania
- United Kingdom (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oxford
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winchester

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Chua L, Friedrich S, Zhang XC. Mirikizumab Pharmacokinetics in Patients with Moderately to Severely Active Ulcerative Colitis: Results from Phase III LUCENT Studies. Clin Pharmacokinet. 2023 Oct;62(10):1479-1491. doi: 10.1007/s40262-023-01281-z. Epub 2023 Aug 23. PMID 37610533
- [Derived] Johnson T, Steere B, Zhang P, Zang Y, Higgs R, Milch C, Reinisch W, Panes J, Huang K, D'Haens G, Krishnan V. Mirikizumab-Induced Transcriptome Changes in Ulcerative Colitis Patient Biopsies at Week 12 Are Maintained Through Week 52. Clin Transl Gastroenterol. 2023 Nov 1;14(11):e00630. doi: 10.14309/ctg.0000000000000630. PMID 37594044
- [Derived] Steere B, Schmitz J, Powell N, Higgs R, Gottlieb K, Liu Y, Jia B, Tuttle JL, Sandborn WJ, Sands BE, D'Haens G, Reinisch W, Krishnan V. Mirikizumab Regulates Genes Involved in Ulcerative Colitis Disease Activity and Anti-TNF Resistance: Results From a Phase 2 Study. Clin Transl Gastroenterol. 2023 Jul 1;14(7):e00578. doi: 10.14309/ctg.0000000000000578. PMID 36881820
- [Derived] Dubinsky MC, Panaccione R, Lewis JD, Sands BE, Hibi T, Lee SD, Naegeli AN, Shan M, Green LA, Morris N, Arora V, Bleakman AP, Belin R, Travis S. Impact of Bowel Urgency on Quality of Life and Clinical Outcomes in Patients With Ulcerative Colitis. Crohns Colitis 360. 2022 Jun 3;4(3):otac016. doi: 10.1093/crocol/otac016. eCollection 2022 Jul. PMID 36777426
- [Derived] Sandborn WJ, Ferrante M, Bhandari BR, Berliba E, Hibi T, D'Haens GR, Tuttle JL, Krueger K, Friedrich S, Durante M, Arora V, Naegeli AN, Schmitz J, Feagan BG. Efficacy and Safety of Continued Treatment With Mirikizumab in a Phase 2 Trial of Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2022 Jan;20(1):105-115.e14. doi: 10.1016/j.cgh.2020.09.028. Epub 2020 Sep 18. PMID 32950748
- [Derived] Sandborn WJ, Ferrante M, Bhandari BR, Berliba E, Feagan BG, Hibi T, Tuttle JL, Klekotka P, Friedrich S, Durante M, Morgan-Cox M, Laskowski J, Schmitz J, D'Haens GR. Efficacy and Safety of Mirikizumab in a Randomized Phase 2 Study of Patients With Ulcerative Colitis. Gastroenterology. 2020 Feb;158(3):537-549.e10. doi: 10.1053/j.gastro.2019.08.043. Epub 2019 Sep 4. PMID 31493397
- See also: Click here for more information about this study: A Study of LY3074828 in Participants With Moderate to Severe Ulcerative Colitis — http://www.lillytrialguide.com/EN-us/studies/colitis/amac

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction: Placebo IV Q4W: Placebo administered every 4 weeks (Q4W) intravenously (IV) during the induction period.
- Induction: 50 mg Mirikizumab IV Q4W: 50 mg mirikizumab administered every 4 weeks (Q4W) intravenously (IV) during the induction period.
  Participants who do not have a clinical response may choose to participate in the unblinded study extension period.
- Induction: 200 mg Mirikizumab IV Q4W: 200 mg mirikizumab administered every 4 weeks (Q4W) intravenously (IV) during the induction period.
  Participants who do not have a clinical response may choose to participate in the unblinded study extension period.
- Induction: 600 mg Mirikizumab IV Q4W: 600 mg mirikizumab administered every 4 weeks (Q4W) intravenously (IV) during the induction period.
  Participants who do not have a clinical response may choose to participate in the unblinded study extension period.
- Maintenance: Placebo SC Q4W: Induction placebo responders: Placebo administered subcutaneously (SC) Q4W during the maintenance period.
- Maintenance: 200 mg Mirikizumab SC Q4W: Induction mirikizumab responders were re-randomized: 200 mg mirikizumab administered subcutaneously (SC) Q4W during the maintenance period.
- Maintenance: 200 mg Mirikizumab SC Q12W: Induction mirikizumab responders were re-randomized: 200 mg mirikizumab administered subcutaneously (SC) once every 12 weeks (Q12W) during the maintenance period.
- Induction Extension: 600mg Mirikizumab IV Q4W: Induction non-responders: 600 mg mirikizumab administered intravenously (IV) once every 4 weeks (Q4W) during the Extension Open-Label.
- Induction Extension: 1000mg Mirikizumab IV Q4W: Induction non-responders: 1000 mg mirikizumab administered intravenously (IV) once every 4 weeks (Q4W) during the Extension Open-Label.
- Maintenance Extension: 200mg Mirikizumab SC Q4W: Extension Induction responders: 200 mg mirikizumab administered subcutaneously (SC) once every 4 weeks (Q4W) during the Extension Open-Label.
Period: Induction Period
Arm/Group | Induction: Placebo IV Q4W | Induction: 50 mg Mirikizumab IV Q4W | Induction: 200 mg Mirikizumab IV Q4W | Induction: 600 mg Mirikizumab IV Q4W | Maintenance: Placebo SC Q4W | Maintenance: 200 mg Mirikizumab SC Q4W | Maintenance: 200 mg Mirikizumab SC Q12W | Induction Extension: 600mg Mirikizumab IV Q4W | Induction Extension: 1000mg Mirikizumab IV Q4W | Maintenance Extension: 200mg Mirikizumab SC Q4W
Started | 63 | 63 | 62 | 61 | 0 (Participants were assigned to this arm during maintenance period.) | 0 (Participants were assigned to this arm during maintenance period.) | 0 (Participants were assigned to this arm during maintenance period.) | 0 | 0 | 0
Received at Least One Dose of Study Drug | 63 | 63 | 62 | 60 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 60 | 61 | 60 | 57 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Did not receive drug | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Period
Arm/Group | Induction: Placebo IV Q4W | Induction: 50 mg Mirikizumab IV Q4W | Induction: 200 mg Mirikizumab IV Q4W | Induction: 600 mg Mirikizumab IV Q4W | Maintenance: Placebo SC Q4W | Maintenance: 200 mg Mirikizumab SC Q4W | Maintenance: 200 mg Mirikizumab SC Q12W | Induction Extension: 600mg Mirikizumab IV Q4W | Induction Extension: 1000mg Mirikizumab IV Q4W | Maintenance Extension: 200mg Mirikizumab SC Q4W
Started | 0 (Participants were assigned to this arm only during induction period.) | 0 (Participants were assigned to this arm only during induction period.) | 0 (Participants were assigned to this arm only during induction period.) | 0 (Participants were assigned to this arm only during induction period.) | 13 (Only participants with a response were re-randomized in maintenance period.) | 47 (Only participants with a response were re-randomized in maintenance period.) | 46 (Only participants with a response were re-randomized in maintenance period.) | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 13 | 47 | 46 | 0 | 0 | 0
Not completed — Rolled Over to Study AMAP (NCT03519945) | 0 | 0 | 0 | 0 | 7 | 41 | 39 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 4 | 2 | 4 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Reason Not Collected | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Period: Induction Extension Period
Arm/Group | Induction: Placebo IV Q4W | Induction: 50 mg Mirikizumab IV Q4W | Induction: 200 mg Mirikizumab IV Q4W | Induction: 600 mg Mirikizumab IV Q4W | Maintenance: Placebo SC Q4W | Maintenance: 200 mg Mirikizumab SC Q4W | Maintenance: 200 mg Mirikizumab SC Q12W | Induction Extension: 600mg Mirikizumab IV Q4W | Induction Extension: 1000mg Mirikizumab IV Q4W | Maintenance Extension: 200mg Mirikizumab SC Q4W
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 32 | 96 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 30 | 84 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 12 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Reason Not Collected | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Maintenance Extension Period
Arm/Group | Induction: Placebo IV Q4W | Induction: 50 mg Mirikizumab IV Q4W | Induction: 200 mg Mirikizumab IV Q4W | Induction: 600 mg Mirikizumab IV Q4W | Maintenance: Placebo SC Q4W | Maintenance: 200 mg Mirikizumab SC Q4W | Maintenance: 200 mg Mirikizumab SC Q12W | Induction Extension: 600mg Mirikizumab IV Q4W | Induction Extension: 1000mg Mirikizumab IV Q4W | Maintenance Extension: 200mg Mirikizumab SC Q4W
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 68
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 68
Not completed — Rolled Over to Study AMAP (NCT03519945) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 57
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Non-responder | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Induction: Placebo IV Q4W: Placebo administered every 4 weeks (Q4W) intravenously (IV).
- Induction: 50 mg Mirikizumab IV Q4W: 50 mg mirikizumab administered every 4 weeks (Q4W) intravenously (IV).
  Participants who do not have a clinical response may choose to participate in the unblinded study extension period.
- Induction: 200 mg Mirikizumab IV Q4W: 200 mg mirikizumab administered every 4 weeks (Q4W) intravenously (IV).
  Participants who do not have a clinical response may choose to participate in the unblinded study extension period.
- Induction: 600 mg Mirikizumab IV Q4W: 600 mg mirikizumab administered every 4 weeks (Q4W) intravenously (IV).
  Participants who do not have a clinical response may choose to participate in the unblinded study extension period.
- Total: Total of all reporting groups
Arm/Group | Induction: Placebo IV Q4W | Induction: 50 mg Mirikizumab IV Q4W | Induction: 200 mg Mirikizumab IV Q4W | Induction: 600 mg Mirikizumab IV Q4W | Total
Number analyzed (Participants) | 63 | 63 | 62 | 61 | 249
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.62 (13.47) | 41.83 (14.06) | 43.35 (14.75) | 42.44 (13.371) | 42.56 (13.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 25 | 23 | 100
  Male | 36 | 38 | 37 | 38 | 149
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 2 | 2 | 7
  Not Hispanic or Latino | 60 | 58 | 59 | 54 | 231
  Unknown or Not Reported | 3 | 2 | 1 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 10 | 5 | 13 | 5 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 5 | 0 | 7
  White | 52 | 57 | 44 | 56 | 209
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Hungary | 5 | 3 | 6 | 4 | 18
  Czechia | 1 | 0 | 0 | 1 | 2
  Japan | 8 | 5 | 13 | 5 | 31
  United Kingdom | 2 | 2 | 0 | 2 | 6
  Moldova | 5 | 7 | 5 | 7 | 24
  Canada | 2 | 1 | 0 | 3 | 6
  Netherlands | 1 | 4 | 4 | 2 | 11
  Belgium | 4 | 7 | 3 | 7 | 21
  Denmark | 0 | 0 | 0 | 1 | 1
  Poland | 15 | 14 | 12 | 8 | 49
  Georgia | 4 | 7 | 2 | 1 | 14
  Lithuania | 4 | 1 | 3 | 1 | 9
  Australia | 1 | 3 | 1 | 2 | 7
  United States | 11 | 9 | 13 | 17 | 50

OUTCOME MEASURES:

1. Primary Outcome: Induction Period: Percentage of Participants With Clinical Remission at Week 12
Description: Clinical remission at week 12 is a defined as achieving a 9-pt Mayo subscore for rectal bleeding=0, stool frequency=0 or 1 with ≥ 1 point decrease from baseline, and endoscopy=0 or 1, excluding Physician's Global Assessment (PGA).
  * Stool Frequency Subscore, based on the participant's diary and scored from 0 (normal number of stools) to 3 (5 or more stools than normal);
  * Rectal Bleeding Subscore, based on the participant's diary and scored from 0 (no blood) to 3 (blood only passed);
  * Endoscopy Subscore, based on colonoscopy or sigmoidoscopy and scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration);
  * Physician's Global Assessment subscore, based on the physician's overall assessment, and scored from 0 (normal) to 3 (severe disease).
  The total score ranges from 0 to 9 points, with higher scores representing more severe disease.
Time Frame: Week 12
Population: Induction Period: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo IV Q4W: Placebo administered every 4 weeks (Q4W) intravenously (IV).
- 50 mg Mirikizumab IV Q4W: 50 mg mirikizumab administered every 4 weeks (Q4W) intravenously (IV).
  Participants who do not have a clinical response may choose to participate in the unblinded study extension period.
- 200 mg Mirikizumab IV Q4W: 200 mg mirikizumab administered every 4 weeks (Q4W) intravenously (IV).
  Participants who do not have a clinical response may choose to participate in the unblinded study extension period.
- 600 mg Mirikizumab IV Q4W: 600 mg mirikizumab administered every 4 weeks (Q4W) intravenously (IV).
  Participants who do not have a clinical response may choose to participate in the unblinded study extension period.
Arm/Group | Placebo IV Q4W | 50 mg Mirikizumab IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 63 | 63 | 62 | 61
percentage of participants | 4.8 [0.0 to 10.0] | 15.9 [6.8 to 24.9] | 22.6 [12.2 to 33.0] | 11.5 [3.5 to 19.5]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 600 mg Mirikizumab IV Q4W; Test type: Superiority; Odds Ratio (OR) = 2.93, 95% CI 2-sided [0.70 to 12.27]
Statistical Analysis 2: Comparison: Placebo IV Q4W vs 200 mg Mirikizumab IV Q4W; Test type: Superiority; Odds Ratio (OR) = 7.22, 95% CI 2-sided [1.88 to 27.65]
Statistical Analysis 3: Comparison: Placebo IV Q4W vs 50 mg Mirikizumab IV Q4W; Test type: Superiority; Odds Ratio (OR) = 3.61, 95% CI 2-sided [0.92 to 14.17]

2. Secondary Outcome: Induction Period: Percentage of Participants With Clinical Response at Week 12
Description: Clinical response at week 12 is defined as a decrease in the 9-point Mayo subscores (rectal bleeding, stool frequency and the endoscopic findings) inclusive of >= 2 points and >=35% from baseline with either a decrease of rectal bleeding subscore of >=1 or rectal bleeding subscore of 0 or 1.
  The Mayo score is a composite score of ulcerative colitis disease activity calculated as the sum of four subscores:
  * Stool Frequency Subscore, based on the participant's diary and scored from 0 (normal number of stools) to 3 (5 or more stools than normal);
  * Rectal Bleeding Subscore, based on the participant's diary and scored from 0 (no blood) to 3 (blood only passed);
  * Endoscopy Subscore, based on colonoscopy or sigmoidoscopy and scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration).
  The total score ranges from 0 to 9 points, with higher scores representing more severe disease.
Time Frame: Week 12
Population: Induction Period: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV Q4W | 50 mg Mirikizumab IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 63 | 63 | 62 | 61
percentage of participants | 20.6 [10.6 to 30.6] | 41.3 [29.1 to 53.4] | 59.7 [47.5 to 71.9] | 49.2 [36.6 to 61.7]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 600 mg Mirikizumab IV Q4W; Test type: Superiority; Odds Ratio (OR) = 3.95, 95% CI 2-sided [1.73 to 8.98]
Statistical Analysis 2: Comparison: Placebo IV Q4W vs 200 mg Mirikizumab IV Q4W; Test type: Superiority; Odds Ratio (OR) = 6.78, 95% CI 2-sided [2.94 to 15.63]
Statistical Analysis 3: Comparison: Placebo IV Q4W vs 50 mg Mirikizumab IV Q4W; Test type: Superiority; Odds Ratio (OR) = 2.78, 95% CI 2-sided [1.23 to 6.29]

3. Secondary Outcome: Induction Period: Percentage of Participants With Endoscopic Remission at Week 12
Description: Endoscopic remission at week 12 is defined as achieving a Mayo endoscopic score of 0 at Week 12. Endoscopy Subscore is based on colonoscopy or sigmoidoscopy and scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration);
  The total score ranges from 0 to 3 points, with higher scores representing more severe disease.
Time Frame: Week 12
Population: Induction Period: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV Q4W | 50 mg Mirikizumab IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 63 | 63 | 62 | 61
percentage of participants | 1.6 [0.0 to 4.7] | 3.2 [0.0 to 7.5] | 3.2 [0.0 to 7.6] | 1.6 [0.0 to 4.8]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 600 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.986, Mantel Haenszel
Statistical Analysis 2: Comparison: Placebo IV Q4W vs 200 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.553, Mantel Haenszel
Statistical Analysis 3: Comparison: Placebo IV Q4W vs 50 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.560, Mantel Haenszel

4. Secondary Outcome: Maintenance Period: Percentage of Participants With Endoscopic Remission at Week 52
Description: Endoscopic remission at week 52 is defined as achieving a Mayo endoscopic subscore of 0 at Week 52. Endoscopy Subscore is based on colonoscopy or sigmoidoscopy and scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration);
  The total score ranges from 0 to 3 points, with higher scores representing more severe disease.
Time Frame: Week 52
Population: Maintenance period: All randomized participants in maintenance period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo SC Q4W: Placebo administered subcutaneously (SC) Q4W during the maintenance period.
- 200 mg Mirikizumab SC Q4W: 200 mg mirikizumab administered subcutaneously (SC) Q4W during the maintenance period.
- 200 mg Mirikizumab SC Q12W: 200 mg mirikizumab administered subcutaneously (SC) once every 12 weeks (Q12W) during the maintenance period
Arm/Group | Placebo SC Q4W | 200 mg Mirikizumab SC Q4W | 200 mg Mirikizumab SC Q12W
Number analyzed (Participants) | 13 | 47 | 46
percentage of participants | 7.7 [0.0 to 22.2] | 14.9 [4.7 to 25.1] | 28.3 [15.2 to 41.3]
Statistical Analysis 1: Comparison: 200 mg Mirikizumab SC Q4W vs 200 mg Mirikizumab SC Q12W; Test type: Superiority; Odds Ratio (OR) = 2.29, 95% CI 2-sided [0.80 to 6.55]

5. Secondary Outcome: Induction Period: Change From Baseline to Week 12 in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score
Description: The IBDQ is a 32-item subject-completed questionnaire that measures 4 aspects of subjects' lives: symptoms directly related to the primary bowel disturbance, systemic symptoms, emotional function, and social function (Guyatt et al. 1989). Responses are graded on a 7-point. Likert scale in which 7 denotes "not a problem at all" and 1 denotes "a very severe problem." Scores range from 32 to 224; a higher score indicates a better quality of life. LS Mean was calculated using MMRM model for post-baseline measures: Variable = Baseline + Geographical Region + Prior Biologic Therapy Group (N) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 12
Population: Induction Period: All randomized participants who had a baseline and at least one post-baseline IBDQ value.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo IV Q4W | 50 mg Mirikizumab IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 60 | 60 | 60 | 56
score on a scale | 22.3 (4.41) | 33.0 (4.52) | 42.8 (4.40) | 45.2 (4.54)
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 600 mg Mirikizumab IV Q4W; Test type: Superiority; Mean Difference (Final Values) = 22.9, 95% CI 2-sided [11.0 to 34.9]
Statistical Analysis 2: Comparison: Placebo IV Q4W vs 200 mg Mirikizumab IV Q4W; Test type: Superiority; Mean Difference (Final Values) = 20.5, 95% CI 2-sided [8.7 to 32.3]
Statistical Analysis 3: Comparison: Placebo IV Q4W vs 50 mg Mirikizumab IV Q4W; Test type: Superiority; Mean Difference (Final Values) = 10.7, 95% CI 2-sided [-1.0 to 22.5]

6. Secondary Outcome: Induction Period: Change From Baseline to Week 12 in 36-Item Short Form Health Survey (SF-36)
Description: SF-36 Health Status Survey is a generic, health-related scale assessing participant's quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health. Domain scores: general health (range: 5-25); physical functioning (range: 10-30); role-physical (range: 4-8); role-emotional (range: 3-15); social functioning (range: 2-10); bodily pain (range: 2-12); vitality (range: 4-20); mental health (range: 5-25). Each raw scale score was converted to a scale score ranging from 0-100 points, with higher values representing a better outcome [(Raw score) - min{raw score}] / (max {raw score} - min{raw score}) x 100]. LS Mean was calculated using Mixed effect Model Repeat Measurement (MMRM) model for post-baseline measures: Variable = Baseline + Geographical Region + Prior Biologic Therapy Group (N) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 12
Population: Induction Period: All randomized participants who had a baseline and at least one post-baseline SF-36 value.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo IV Q4W | 50 mg Mirikizumab IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 60 | 60 | 60 | 56
score on a scale
  Physical Component Score: number analyzed (Participants) | 60 | 60 | 59 | 56
  Physical Component Score | 3.4 (0.83) | 6.2 (0.86) | 5.9 (0.83) | 6.9 (0.85)
  Mental Component Score | 3.2 (1.22) | 4.5 (1.26) | 6.8 (1.20) | 8.8 (1.25)
  Physical Functioning: number analyzed (Participants) | 60 | 60 | 59 | 56
  Physical Functioning | 2.1 (0.76) | 3.7 (0.78) | 4.6 (0.74) | 6.2 (0.77)
  Role-Physical | 4.5 (1.19) | 7.5 (1.22) | 7.2 (1.17) | 8.0 (1.22)
  Bodily Pain | 3.7 (1.15) | 7.9 (1.18) | 8.9 (1.14) | 10.0 (1.18)
  General Health | 3.1 (0.93) | 3.8 (0.96) | 4.3 (0.92) | 5.1 (0.96)
  Vitality | 3.3 (1.25) | 6.5 (1.28) | 7.5 (1.23) | 9.7 (1.28)
  Social Functioning | 6.5 (1.22) | 8.0 (1.26) | 9.4 (1.21) | 11.6 (1.26)
  Role-Emotional | 3.0 (1.22) | 3.7 (1.26) | 5.5 (1.20) | 7.6 (1.25)
  Mental Health | 1.9 (1.18) | 3.7 (1.22) | 6.4 (1.17) | 7.6 (1.21)

7. Secondary Outcome: Induction Period: Change From Baseline to Week 12 in Patient's Global Impressions of Severity (PGI-S) Score
Description: PGI-S is a 1-item subject-rated questionnaire designed to assess the subject's impression of their disease symptoms at baseline (Guy 1976; Yalcin and Bump 2003). Responses are graded on a 7-point scale in which a score of 1 indicates that the subject's symptom(s) are "normal," a score of 2 indicates that the subject feels "borderline ill," a score of 3 indicates that the subject feels "mildly ill," a score of 4 indicates that the subject(s) feel "moderately ill," and scores of 5, 6, and 7 indicate that the subject feels "markedly ill," "severely ill," and "extremely ill," respectively. LS Mean was calculated using MMRM model for post-baseline measures: Variable = Baseline + Geographical Region + Prior Biologic Therapy Group (N) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 12
Population: Induction Period: All randomized participants who had a baseline and at least one post-baseline PGI-S value.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo IV Q4W | 50 mg Mirikizumab IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 60 | 60 | 60 | 56
score on a scale | -0.84 (0.19) | -1.43 (0.20) | -1.90 (0.18) | -1.74 (0.19)
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 600 mg Mirikizumab IV Q4W; Test type: Superiority; Mean Difference (Final Values) = -0.90, 95% CI 2-sided [-1.39 to -0.41]
Statistical Analysis 2: Comparison: Placebo IV Q4W vs 200 mg Mirikizumab IV Q4W; Test type: Superiority; Mean Difference (Final Values) = -1.06, 95% CI 2-sided [-1.54 to -0.59]
Statistical Analysis 3: Comparison: Placebo IV Q4W vs 50 mg Mirikizumab IV Q4W; Test type: Superiority; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-1.07 to -0.11]

8. Secondary Outcome: Induction Period: Patient's Global Impressions of Improvement (PGI-I) Score at Week 12
Description: PGI-I scale is a subject-rated instrument designed to assess the subject's impression of change in their symptom(s) (Guy 1976; Yalcin and Bump 2003). Responses are graded on a 7-point Likert scale in which a score of 1 indicates that the subject's symptom(s) is "very much better," a score of 4 indicates that the subject's symptom(s) has experienced "no change," and a score of 7 indicates that the subject's symptom(s) is "very much worse."
Time Frame: Week 12
Population: Induction Period: All randomized participants who had a baseline and at least one post-baseline PGI-I value.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo IV Q4W | 50 mg Mirikizumab IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 63 | 62 | 61 | 60
score on a scale | 3.37 (1.46) | 2.69 (1.31) | 2.39 (0.99) | 2.53 (1.16)

9. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration-Time Curve During Dosing Interval at Steady State (AUCss, Tau) of Mirikizumab
Description: Pharmacokinetics (PK): Area Under the Concentration-Time Curve During Dosing Interval at Steady State (AUCss, tau) of Mirikizumab
Time Frame: Induction Period: Day (D) 1, D15 ± 2d, D29 ± 2d, D43 ± 2d, D57 ± 2d, D78-85; Maintenance Period: D85-92,D113± 7d,D141± 7d,D169± 7d,D225 ±7d,D281 ±7d,D337 ±7d,D393± 7d,D448± 7d,D504± 7d,D560± 7d,D616± 7d,D672± 7d,D728± 7d,D784± 7d,D840± 7d
Population: All participants who received at least one dose of mirikizumab in the induction and maintenance period who had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*hour/milligram(ug*hr/ml)
Groups:
- 50 mg Mirikizumab IV Q4W: 50 mg mirikizumab administered every 4 weeks (Q4W) intravenously (IV) during the induction period. Participants who do not have a clinical response may choose to participate in the unblinded study extension period.
- 200 mg Mirikizumab IV Q4W: 200 mg mirikizumab administered every 4 weeks (Q4W) intravenously (IV) during the induction period.
  Participants who do not have a clinical response may choose to participate in the unblinded study extension period.
- 600 mg Mirikizumab IV Q4W: 600 mg mirikizumab administered every 4 weeks (Q4W) intravenously (IV) during the induction period.
  Participants who do not have a clinical response may choose to participate in the unblinded study extension period.
Arm/Group | 50 mg Mirikizumab IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W | 200 mg Mirikizumab SC Q4W | 200 mg Mirikizumab SC Q12W
Number analyzed (Participants) | 63 | 62 | 61 | 47 | 46
Microgram*hour/milligram(ug*hr/ml) | 3330 (42.5) | 10100 (35.0) | 24900 (36.6) | 3700 (41.5) | 1270 (42.3)

10. Secondary Outcome: Induction Period: Percentage of Participants With Symptomatic Remission at Week 12
Description: Symptomatic remission is defined as a stool frequency score of 0 or 1 and a rectal bleeding score of 0.
  * Stool Frequency Subscore is based on the participant's diary and scored from 0 (normal number of stools) to 3 (5 or more stools than normal).
  * Rectal Bleeding Subscore is based on the participant's diary and scored from 0 (no blood) to 3 (blood only passed).
  The total score ranges from 0 to 1 points, with higher scores representing more severe disease.
  The percentage of response is calculated by dividing number of participants in the specified category by number of participants with non-missing values multiplied by 100.
Time Frame: Week 12
Population: Induction Period: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV Q4W | 50 mg Mirikizumab IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 63 | 63 | 62 | 61
percentage of participants | 20.6 [10.6 to 30.6] | 36.5 [24.6 to 48.4] | 58.1 [45.8 to 70.3] | 45.9 [33.4 to 58.4]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 600 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 3.61, 95% CI 2-sided [1.57 to 8.31]
Statistical Analysis 2: Comparison: Placebo IV Q4W vs 200 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.54, 95% CI 2-sided [2.81 to 15.20]
Statistical Analysis 3: Comparison: Placebo IV Q4W vs 50 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.054, Regression, Logistic; Odds Ratio (OR) = 2.27, 95% CI 2-sided [0.98 to 5.22]

11. Secondary Outcome: Maintenance Period: Percentage of Participants With Symptomatic Remission at Week 52
Description: Symptomatic remission is defined as a stool frequency score of 0 or 1 and a rectal bleeding score of 0.
  * Stool Frequency Subscore , based on the participant's diary and scored from 0 (normal number of stools) to 3 (5 or more stools than normal);
  * Rectal Bleeding Subscore , based on the participant's diary and scored from 0 (no blood) to 3 (blood only passed);
  * Endoscopy Subscore , based on colonoscopy or sigmoidoscopy and scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration);
  * Physician's Global Assessment subscore, based on the physician's overall assessment, and scored from zero (normal) to 3 (severe disease).
  The total score ranges from 0 to 1 points, with higher scores representing more severe disease.
  The percentage of response is calculated by dividing number of participants in the specified category by number of participants with non-missing values multiplied by 100.
Time Frame: Week 52
Population: Maintenance period: All randomized participants in maintenance period.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo SC Q4W | 200 mg Mirikizumab SC Q4W | 200 mg Mirikizumab SC Q12W
Number analyzed (Participants) | 13 | 47 | 46
Percentage of Participants | 53.8 [26.7 to 80.9] | 76.6 [64.5 to 88.7] | 65.2 [51.5 to 79.0]
Statistical Analysis 1: Comparison: 200 mg Mirikizumab SC Q4W vs 200 mg Mirikizumab SC Q12W; Test type: Superiority; p = 0.131, Regression, Logistic; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.19 to 1.24]

12. Secondary Outcome: Induction Period: Percentage of Participants With Endoscopic Improvement at Week 12
Description: Endoscopic Improvement defined as achieving an endoscopic findings subscore of 0 or 1. Endoscopy Subscore is based on colonoscopy or sigmoidoscopy and scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration). The percentage of response is calculated by dividing number of participants in the specified category by number of participants with non-missing values multiplied by 100.
Time Frame: Week 12
Population: Induction Period: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV Q4W | 50 mg Mirikizumab IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 63 | 63 | 62 | 61
percentage of participants | 6.3 [0.3 to 12.4] | 23.8 [13.3 to 34.3] | 30.6 [19.2 to 42.1] | 13.1 [4.6 to 21.6]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 600 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.215, Regression, Logistic; Odds Ratio (OR) = 2.25, 95% CI 2-sided [0.63 to 8.07]
Statistical Analysis 2: Comparison: Placebo IV Q4W vs 200 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.70, 95% CI 2-sided [2.37 to 25.00]
Statistical Analysis 3: Comparison: Placebo IV Q4W vs 50 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.012, Regression, Logistic; Odds Ratio (OR) = 4.62, 95% CI 2-sided [1.41 to 15.14]

13. Secondary Outcome: Maintenance Period: Percentage of Participants With Endoscopic Improvement at Week 52
Description: as for outcome 12
Time Frame: Week 52
Population: Maintenance period: All randomized participants in maintenance period.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Placebo SC Q4W | 200 mg Mirikizumab SC Q4W | 200 mg Mirikizumab SC Q12W
Number analyzed (Participants) | 13 | 47 | 46
Percentage of Participants | 15.4 [0.0 to 35.0] | 57.4 [43.3 to 71.6] | 47.8 [33.4 to 62.3]
Statistical Analysis 1: Comparison: 200 mg Mirikizumab SC Q4W vs 200 mg Mirikizumab SC Q12W; Test type: Superiority; p = 0.428, Regression, Logistic; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.31 to 1.65]

ADVERSE EVENTS:
Time Frame: Up To 39 Months
Description: All participants who received at least one dose of study. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- Induction: 50 mg Mirikizumab Administered Every 4 Weeks (Q4W): 50 mg mirikizumab administered every 4 weeks (Q4W) intravenously (IV) during the induction period.
  Participants who do not have a clinical response may choose to participate in the unblinded study extension period.
- Maintenance: 200 mg Mirikizumab SC Q4W: Induction mirikizumab responders: 200 mg mirikizumab administered subcutaneously (SC) Q4W during the maintenance period.
- Maintenance: 200 mg Mirikizumab SC Q12W: Induction mirikizumab responders: 200 mg mirikizumab administered subcutaneously (SC) once every 12 weeks (Q12W) during the maintenance period.
- Induction Extension:1000mg Mirikizumab IV Q4W: Induction non-responders: 1000 mg mirikizumab administered intravenously (IV) ) once every 4 weeks (Q4W) during the Extension Open-Label.
Arm/Group | Induction: Placebo IV Q4W | Induction: 50 mg Mirikizumab Administered Every 4 Weeks (Q4W) | Induction: 200 mg Mirikizumab IV Q4W | Induction: 600 mg Mirikizumab IV Q4W | Maintenance: Placebo SC Q4W | Maintenance: 200 mg Mirikizumab SC Q4W | Maintenance: 200 mg Mirikizumab SC Q12W | Induction Extension: 600mg Mirikizumab IV Q4W | Induction Extension:1000mg Mirikizumab IV Q4W | Maintenance Extension: 200mg Mirikizumab SC Q4W
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63 | 0/62 | 0/60 | 0/13 | 0/47 | 0/46 | 0/32 | 0/96 | 0/68
Serious Adverse Events (participants affected / at risk) | 2/63 | 0/63 | 2/62 | 3/60 | 2/13 | 2/47 | 1/46 | 1/32 | 5/96 | 3/68
Other Adverse Events (participants affected / at risk) | 18/63 | 14/63 | 8/62 | 14/60 | 11/13 | 27/47 | 30/46 | 9/32 | 8/96 | 30/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction: Placebo IV Q4W (N=63) | Induction: 50 mg Mirikizumab Administered Every 4 Weeks (Q4W) (N=63) | Induction: 200 mg Mirikizumab IV Q4W (N=62) | Induction: 600 mg Mirikizumab IV Q4W (N=60) | Maintenance: Placebo SC Q4W (N=13) | Maintenance: 200 mg Mirikizumab SC Q4W (N=47) | Maintenance: 200 mg Mirikizumab SC Q12W (N=46) | Induction Extension: 600mg Mirikizumab IV Q4W (N=32) | Induction Extension:1000mg Mirikizumab IV Q4W (N=96) | Maintenance Extension: 200mg Mirikizumab SC Q4W (N=68)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug dependence (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Induction: Placebo IV Q4W (N=63) | Induction: 50 mg Mirikizumab Administered Every 4 Weeks (Q4W) (N=63) | Induction: 200 mg Mirikizumab IV Q4W (N=62) | Induction: 600 mg Mirikizumab IV Q4W (N=60) | Maintenance: Placebo SC Q4W (N=13) | Maintenance: 200 mg Mirikizumab SC Q4W (N=47) | Maintenance: 200 mg Mirikizumab SC Q12W (N=46) | Induction Extension: 600mg Mirikizumab IV Q4W (N=32) | Induction Extension:1000mg Mirikizumab IV Q4W (N=96) | Maintenance Extension: 200mg Mirikizumab SC Q4W (N=68)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Colitis ulcerative (Gastrointestinal disorders) | 6 (6) | 2 (2) | 1 (1) | 1 (1) | 7 (10) | 4 (4) | 7 (7) | 0 (0) | 0 (0) | 7 (7)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (14) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 4 (5) | 3 (3) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (7) | 5 (5) | 3 (3) | 5 (5) | 1 (2) | 6 (12) | 8 (10) | 5 (5) | 7 (8) | 14 (21)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 4 (8)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 5 (7) | 3 (3) | 0 (0) | 0 (0) | 6 (7)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin b12 decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin d decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 6 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 1 (1) | 4 (5) | 1 (1) | 5 (9) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/27 (0) | 0/25 (0) | 0/25 (0) | 0/22 (0) | 1/5 (1) | 0/20 (0) | 0/24 (0) | 0/12 (0) | 0/33 (0) | 0/25 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT02589665/SAP_000.pdf
  • Study Protocol (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT02589665/Prot_001.pdf